CLINICAL TRIAL: NCT01879280
Title: Effect of Craniotomy on Temporalis Function
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Kyle Weaver, Assistant Professor Neurological Surgery, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 100387
Record Dates: First submitted 2010-04-29; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Pterional Craniotomy
Keywords: pterional craniotomy; osteoplastic craniotomy; temporalis; minimally-invasive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- osteoplastic craniotomy (Experimental): Half of the study population will be randomized to traditional pterional craniotomy as the method of exposure. The other half will be randomized to osteoplastic craniotomy as the method of exposure. All other aspects of medical care will remain the same.
  Interventions: Procedure: Traditional pterional craniotomy; Procedure: Osteoplastic craniotomy
- traditional pterional craniotomy (Active Comparator): traditional pterional craniotomy
  Interventions: Procedure: Traditional pterional craniotomy

INTERVENTIONS:
Procedure: Traditional pterional craniotomy — In the standard pterional craniotomy group, the attachment of the temporalis will be cut and the temporalis will be mobilized prior to exposure of the underlying bony calvarium. This maneuver is currently accepted for use by the majority of neurosurgeons nationwide.
Procedure: Osteoplastic craniotomy — In the osteoplastic group, the temporalis will be left attached to the bony calvarium prior to exposure of the tumor. There are ways to turn a bone flap with the temporalis still attached (i.e., an "osteoplastic craniotomy"). However, this method is thought to be slightly more time-consuming and is used less often in many centers. Aside from the extra time involved, we do not feel that leaving the temporalis attached to the bony calvarium disadvantages the patient in any fashion and may--in fact--result in less post-operative morbidity.
  Arms: osteoplastic craniotomy

SUMMARY:
The scientific objectives of this study are to systematically study the problems that are created by incising the attachment of the temporalis muscle in a randomized group of patients, and to determine whether another approach that does not detach the temporalis muscle results in less post-operative morbidity. Cutting through the attachment of the temporalis muscle to the skull is a widely-accepted procedure used to gain access to the skull prior to the drilling used for a pterional craniotomy (one of the most frequent types of surgeries used in neurosurgical practice). Despite the frequent use of this maneuver and the known sequelae of temporalis mobilization (e.g. post-operative myofascial pain, temporalis weakness, and pain with mastication), very little is known about the true incidence of these post-operative symptoms. Furthermore, there is very little objective evidence at the present time to support the claim that the incidence and severity of these post-operative phenomena can be decreased with use of an osteoplastic craniotomy (a procedure where the temporalis is left attached to the bony calvarium). The investigators would like to evaluate whether this slightly more time-consuming and technically demanding approach is less morbid in this respect than the contemporary pterional approach. Special note is made that the osteoplastic approach has been used in standard neurosurgical practice for quite some time.

DETAILED DESCRIPTION:
In contemporary neurosurgery, when performing a pterional craniotomy, neurosurgeons have been taught to cut through and detach the temporalis before drilling the skull to "turn a bone flap". While there are ways to turn a bone flap with the temporalis still attached (i.e., an "osteoplastic craniotomy"), this is thought to be slightly more time-consuming and is used less often in many centers. Additionally, there is a common misconception that osteoplastic craniotomy does not allow an equivalent view, although recent evidence suggests that the surgical exposure in the two approaches is no different. Aside from the extra time involved, we do not feel that leaving the temporalis attached to the bony calvarium disadvantages the patient in any fashion (and-in fact-may result in less post-operative morbidity). We are interested in this project because there is actually very little objective data regarding the morbidity people experience when the temporalis muscle is cut and mobilized prior to drilling the skull. If, in this study, we find that the group randomized to traditional pterional craniotomy experiences significantly more morbidity than the group randomized to osteoplastic craniotomy, this may justify conversion to an osteoplastic craniotomy in many or all instances.

We wish to quantify the morbidity that is associated with the specific methods used to detach the temporalis muscle from the skull. Many variables regarding the way the temporalis is detached will be recorded and assessed in the group randomized to traditional pterional craniotomy. Additionally, many methods will be used to measure post-operative temporalis atrophy and/or dysfunction in the two randomized groups. After post-operative morbidity has been quantified, we plan to compare the traditional pterional group to the osteoplastic group and assess for significance.

ELIGIBILITY:
Inclusion Criteria:

* o The selection of participants is based solely on future plans to undergo a pterional craniotomy for resection of a tumor.

Exclusion Criteria:

* o Because patient feedback and participation is necessary, cognitively impaired patients are excluded from this study.

  * Also, generalized cachexia, prior history of craniotomy, or any other reason for baseline temporalis asymmetry or poor wound healing is also reason for exclusion from this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Post-operative mobility of the jaw (e.g. lateral excursion and protrusion) | 6 weeks and 1 year post-operatively
  Data regarding baseline and post-operative range-of-motion of the mouth will be collected before and after surgery.

SECONDARY OUTCOMES:
Post-operative pain with chewing | 6 weeks and 1 year
  Data regarding baseline and post-operative pain with chewing will be obtained at 6 months and 1 year.
Post-operative cosmesis of the temporal region | 6 weeks and 1 year post-operatively
  Data regarding baseline and post-operative cosmesis will be obtained and 6 weeks and 1 year post-operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Univesity Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Balasingam V, Noguchi A, McMenomey SO, Delashaw JB Jr. Modified osteoplastic orbitozygomatic craniotomy. Technical note. J Neurosurg. 2005 May;102(5):940-4. doi: 10.3171/jns.2005.102.5.0940. PMID 15926727
- [Result] Rocha-Filho PA, Fujarra FJ, Gherpelli JL, Rabello GD, de Siqueira JT. The long-term effect of craniotomy on temporalis muscle function. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Nov;104(5):e17-21. doi: 10.1016/j.tripleo.2007.05.029. Epub 2007 Aug 30. PMID 17764986
- [Result] de Andrade Junior FC, de Andrade FC, de Araujo Filho CM, Carcagnolo Filho J. Dysfunction of the temporalis muscle after pterional craniotomy for intracranial aneurysms. Comparative, prospective and randomized study of one flap versus two flaps dieresis. Arq Neuropsiquiatr. 1998 Jun;56(2):200-5. doi: 10.1590/s0004-282x1998000200006. PMID 9698728
- See also: paper #3 — http://www.ncbi.nlm.nih.gov/pubmed/9698728